CLINICAL TRIAL: NCT05692609
Title: Comparison of the Acoustic Voice Quality of Edentulous Patients Treated With Two-implant Overdentures or All-on-4 Concept
Brief Title: The Effect of Implant-supported Prosthesis on Acoustic Voice Quality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist. Prof., Marmara University
Other Study IDs: MUDHF_PTT_02
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Edentulous Jaw
Keywords: Dental Prosthesis, Implant-Supported; Speech Acoustics
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Implant overdenture group: In the control session, participants' acoustic sound quality, implant and prosthesis success will be measured.
- All-on-4 group: In the control session, participants' acoustic sound quality, implant and prosthesis success will be measured.

SUMMARY:
The primary aim of this study was to compare the acoustic sound quality of edentulous patients rehabilitated with two-implant overdentures or the all-on-4 concept. The secondary aims were to evaluate the effect of implant and prosthetic success on acoustics.

ELIGIBILITY:
Inclusion Criteria:

* No voice disorder or speech therapy
* The implant prosthesis was made at least one year ago, delivered to the patient, and continues to be used

Exclusion Criteria:

* Smoking (>10 cigarettes/day) or substance use
* History of acute or chronic respiratory diseases
* Overdenture prosthesis on three or 4 implants
* History of speech and hearing problems
* Patients who have lost any implants before the control

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with all-on-4 or two-implant overdentures whose surgery and prosthesis were performed at Marmara University Faculty of Dentistry clinics
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Acoustic voice quality index | At the follow-up session (approximately one year after delivery of the prosthesis)
  The acoustic Voice Quality Index (AVQI) measures the perceived quality of a voice signal. It is based on evaluating several acoustic parameters that are known to be related to the perceived quality of speech. These parameters include measures of loudness, pitch, and spectral tilt, as well as measures of the presence of noise and other distortions in the signal. Acoustic voice quality will be evaluated in accordance with the AVQI index. During the control session, two separate voice recordings will be made with and without the participants' dentures in the mouth and transferred to the software. The score obtained according to the AVQI index will be used for statistical analysis between groups.

SECONDARY OUTCOMES:
Implant success | At the follow-up session (approximately one year after delivery of the prosthesis)
  Implant success will be defined according to the following criteria:
  * Clinical stability and immobility (0); (1)
  * Full functionality (0); (1)
  * Absence of pain on mild percussion (0); (1)
  * Healthy peri-implant soft tissue and radiolucency at probing (0); (1)
  * Absence of other radiographic pathologic conditions (0); (1). Implant loss and implant mobility will be recorded on standardized documentation forms, as will complications related to prostheses.
Prosthetic Success | At the follow-up session (approximately one year after delivery of the prosthesis)
  The success of the prosthetic treatment will be evaluated according to the criteria set by Awad and Feine. Participants will be asked about their overall satisfaction with their prosthesis. Also;
  * Prosthesis stability (0) - (10)
  * Comfort (0) - (10)
  * Chewing skills (0) - (10)
  * Speaking skills (0) - (10)
  * Ease of cleaning (0) - (10) and
  * They will be asked to rate their aesthetic appearance (Awad & Feine, 1998).
  Participants will rate each item on a 10 cm visual analog scale, where the anchor words are "not at all satisfied" for zero and "completely satisfied" for 10. Participants will be asked to draw a vertical line at the point on the scale that best reflects their responses, where higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tyrovolas S, Koyanagi A, Panagiotakos DB, Haro JM, Kassebaum NJ, Chrepa V, Kotsakis GA. Population prevalence of edentulism and its association with depression and self-rated health. Sci Rep. 2016 Nov 17;6:37083. doi: 10.1038/srep37083. PMID 27853193
- [Background] Marcus PA, Joshi A, Jones JA, Morgano SM. Complete edentulism and denture use for elders in New England. J Prosthet Dent. 1996 Sep;76(3):260-6. doi: 10.1016/s0022-3913(96)90169-9. PMID 8887798
- [Background] Romandini M, Baima G, Antonoglou G, Bueno J, Figuero E, Sanz M. Periodontitis, Edentulism, and Risk of Mortality: A Systematic Review with Meta-analyses. J Dent Res. 2021 Jan;100(1):37-49. doi: 10.1177/0022034520952401. Epub 2020 Aug 31. PMID 32866427
- [Background] Nowjack-Raymer RE, Sheiham A. Association of edentulism and diet and nutrition in US adults. J Dent Res. 2003 Feb;82(2):123-6. doi: 10.1177/154405910308200209. PMID 12562885
- [Background] Slade GD, Akinkugbe AA, Sanders AE. Projections of U.S. Edentulism prevalence following 5 decades of decline. J Dent Res. 2014 Oct;93(10):959-65. doi: 10.1177/0022034514546165. Epub 2014 Aug 21. PMID 25146182
- [Background] Douglass CW, Watson AJ. Future needs for fixed and removable partial dentures in the United States. J Prosthet Dent. 2002 Jan;87(1):9-14. doi: 10.1067/mpr.2002.121204. PMID 11807477
- [Background] Malo P, Rangert B, Nobre M. "All-on-Four" immediate-function concept with Branemark System implants for completely edentulous mandibles: a retrospective clinical study. Clin Implant Dent Relat Res. 2003;5 Suppl 1:2-9. doi: 10.1111/j.1708-8208.2003.tb00010.x. PMID 12691645
- [Background] Zitzmann NU, Scharer P, Marinello CP. Factors influencing the success of GBR. Smoking, timing of implant placement, implant location, bone quality and provisional restoration. J Clin Periodontol. 1999 Oct;26(10):673-82. doi: 10.1034/j.1600-051x.1999.261007.x. PMID 10522779
- [Background] Jacobs R, Manders E, Van Looy C, Lembrechts D, Naert I, van Steenberghe D. Evaluation of speech in patients rehabilitated with various oral implant-supported prostheses. Clin Oral Implants Res. 2001 Apr;12(2):167-73. doi: 10.1034/j.1600-0501.2001.012002167.x. PMID 11251667
- [Background] Lu FL, Matteson S. Speech tasks and interrater reliability in perceptual voice evaluation. J Voice. 2014 Nov;28(6):725-32. doi: 10.1016/j.jvoice.2014.01.018. Epub 2014 May 17. PMID 24841668
- [Background] Umapathy K, Krishnan S, Parsa V, Jamieson DG. Discrimination of pathological voices using a time-frequency approach. IEEE Trans Biomed Eng. 2005 Mar;52(3):421-30. doi: 10.1109/TBME.2004.842962. PMID 15759572
- [Background] Asiaee M, Nourbakhsh M, Vahedian-Azimi A, Zare M, Jafari R, Atashi SS, Keramatfar A. The feasibility of using acoustic measures for predicting the Total Opacity Scores of chest computed tomography scans in patients with COVID-19. Clin Linguist Phon. 2024 Mar;38(2):97-115. doi: 10.1080/02699206.2022.2160659. Epub 2023 Jan 2. PMID 36592050
- [Background] Shabnam S, Pushpavathi M, Gopi Sankar R, Sridharan KV, Vasanthalakshmi MS. A Comprehensive Application for Grading Severity of Voice Based on Acoustic Voice Quality Index v.02.03. J Voice. 2025 Jan;39(1):287.e1-287.e9. doi: 10.1016/j.jvoice.2022.08.013. Epub 2022 Oct 1. PMID 36192290
- [Background] Barsties V Latoszek B, Ulozaite-Staniene N, Petrauskas T, Uloza V, Maryn Y. Diagnostic Accuracy of Dysphonia Classification of DSI and AVQI. Laryngoscope. 2019 Mar;129(3):692-698. doi: 10.1002/lary.27350. Epub 2018 Sep 10. PMID 30203473
- [Background] Englert M, Barsties V Latoszek B, Maryn Y, Behlau M. Validation of the Acoustic Voice Quality Index, Version 03.01, to the Brazilian Portuguese Language. J Voice. 2021 Jan;35(1):160.e15-160.e21. doi: 10.1016/j.jvoice.2019.07.024. Epub 2019 Aug 29. PMID 31474432
- [Background] Faham M, Laukkanen AM, Ikavalko T, Rantala L, Geneid A, Holmqvist-Jamsen S, Ruusuvirta K, Pirila S. Acoustic Voice Quality Index as a Potential Tool for Voice Screening. J Voice. 2021 Mar;35(2):226-232. doi: 10.1016/j.jvoice.2019.08.017. Epub 2019 Sep 30. PMID 31582330
- [Background] Yesilli-Puzella G, Tadihan-Ozkan E, Maryn Y. Validation and Test-Retest Reliability of Acoustic Voice Quality Index Version 02.06 in the Turkish Language. J Voice. 2022 Sep;36(5):736.e25-736.e32. doi: 10.1016/j.jvoice.2020.08.021. Epub 2020 Sep 20. PMID 32962941